CLINICAL TRIAL: NCT01066078
Title: Echocardiography and PEA Measurements in CRT Therapy
Brief Title: Echocardiography and Peak Endocardial Acceleration (PEA) Measurements in Cardiac Resynchronization Therapy (CRT)
Status: Completed | Type: Observational
Sponsor: LivaNova (Industry)
Responsible Party: Erwan DONAL, CCP, CHU Pontchaillou 35033 RENNES France
Other Study IDs: RGEA01 - CAP PEA; RGEA01
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Congestive Heart Failure
Keywords: heart failure - congestive; Cardiovascular imaging agents/Techniques]; Echocardiography; Other diagnostic testing; Other Treatment; Recipients of cardiac resynchronization therapy systems
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRT recipients
  Interventions: Other: Echocardiography and SonR recording

INTERVENTIONS:
Other: Echocardiography and SonR recording

SUMMARY:
This study used an external endocardial acceleration sensor (sonR sensor), placed on the patient's chest, to time the closure of aortic and mitral valves, and compared its performance with echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Every patient coming in the participating centers for an echocardiographic exam and implanted with a pacemaker or an implantable cardioverter defibrillator (ICD) can be included in the study.

Exclusion Criteria:

* Inability to understand the patient information sheet.
* Minor patient or pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CRT recipients
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The timings of mitral (tMC) and aortic (tAC) valves closure by echocardiography and sonR | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Erwan DONAL, MD, Principal Investigator — CHU Rennes
Locations (4):
- France (4):
  - Nouvelles Cliniques Nantaises, Nantes
  - Clinique Bizet, Paris
  - CHU Pontchaillou, Rennes
  - CHU Rennes, Rennes